CLINICAL TRIAL: NCT03397199
Title: A Phase II Clinical Trial of Apatinib Plus S-1 as the Therapy of Advanced Colorectal Cancer
Brief Title: Study of Apatinib Plus S-1 as the Therapy of Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HNP052
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — apatinib; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib + S-1 (Experimental): Apatinib + S-1
  Interventions: Drug: Apatinib + S-1

INTERVENTIONS:
Drug: Apatinib + S-1 — Apatinib 250mg/d,q.d.,p.o. A course of treatment need 21days. S-1 40-60mg（40mg bid BSA <1.4, 60mg bid BSA>1.4），bid,from day1-day 14.

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Apatinib plus S-1 as the Therapy of Advanced Colorectal Cancer.

DETAILED DESCRIPTION:
Colorectal cancer is a common clinical gastrointestinal cancer. In addition to the early diagnosis of some patients, approximately 50% of patients have had distant metastases at the time of diagnosis. For patients with advanced colorectal cancer, systemic chemotherapy is the main treatment. We consider to add apatinib,a tyrosine kinase inhibitor of VEGF,to the therapy of these patients. We designed the study to explore the possibility of apatinib for Advanced Colorectal Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form prior to patient entry.
2. Histologically or cytologically diagnosed as metastatic colon or rectal adenocarcinoma patients.
3. The second-line standard regimen failed (disease progression) and the chemotherapy regimen included fluorouracil (5-FU / capecitabine / tioguanide), oxaliplatin and irinotecan from the last chemotherapy> 14 days.
4. ≥ 18 and ≤ 70 years of age.
5. Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
6. Life expectancy of more than 3 months.
7. According to the solid tumor efficacy evaluation criteria RECISTv1.1 standards, at least one measurable lesions. If the previous treatment of local treatment (radiotherapy, radiofrequency, intervention, etc.) is the only focus of lesions, the request must have a clear imaging progress.
8. Adequate hepatic, renal, heart, and hematologic functions: ANC ≥1.5×109/L, PLT ≥ 100×109/L, HB ≥ 90 g/L, TBIL ≤ 1.5×ULN, ALT or AST≤ 2.5×ULN (or ≤ 5×ULN in patients with liver metastases), Serum Cr≤ 1.5×ULN, Cr clearance ≥ 60 mL/min.
9. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 6 months after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 6 months after last dose of study drug.

Exclusion Criteria:

1. Uncontrollable hypertension (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg, despite optimal medical therapy).
2. Poor glycemic control in diabetes.
3. Acute cerebral infarction, or recovery period <2 months.
4. A variety of factors that affect oral absorption (such as inability to swallow, nausea, vomiting, chronic diarrhea, intestinal obstruction, etc.).
5. Patients with gastrointestinal bleeding risk may not be included, including the following: (1) active peptic ulcer lesions and fecal occult blood (++); (2) history of melena and vomiting within 3 months；Fecal occult blood (+) is not an exclusion criterion.
6. Coagulation dysfunction (INR> 1.5, PT> ULN + 4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment.
7. Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g.
8. Pregnant or lactating women.
9. Cytotoxic drug treatment, radiotherapy within 2 weeks after treatment; had taken two or more oral targeted drugs.
10. Other malignant tumors, cutaneous basal cell carcinoma, and cervical cancer in situ in the past 5 years.
11. The investigators believe there is any condition that may harm the subject or result in the subject's inability to meet or perform the research requirements
12. Severe liver and kidney dysfunction (grade 4) patients should be excluded.
13. Any allergy to apatinib should be excluded.
14. Persons with a history of substance abuse who can not be abdicated or have mental disorders.
15. Previously used regurgitine is not an exclusion criterion.
16. According to the judgment of the researcher, there is a concomitant disease that seriously endangers the patient's safety or affects the patient in completing the study.
17. Patients who underwent surgery within 4 weeks prior to the start of treatment or who had major trauma or fractures. Or there is an unhealed wound before treatment.
18. Patients with severe heart disease such as grade III or above (NYHA standard) congestive heart failure, grade III or above (CCS standard) angina, or a history of myocardial infarction within 6 months prior to the start of treatment, or patients requiring medication Arrhythmia.
19. A brain metastasis, meningeal transfer.
20. Active HBV infection and refusal of regular antiviral treatment.
21. Active tuberculosis patients.
22. Participate in any drug or medical device clinical trial within 1 month before the test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause
Disease Control Rate (DCR) | up to 1 year
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR
  + PR + SD)
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital; Ning Li, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Li N, Deng W, Zhang G, Du Y, Guo Y, Ma Y, Wei C, Bie L, Zhang C, Song T, Luo S, Fang B. Low-Dose Apatinib Combined With S-1 in Refractory Metastatic Colorectal Cancer: A Phase 2, Multicenter, Single-Arm, Prospective Study. Front Oncol. 2021 Sep 2;11:728854. doi: 10.3389/fonc.2021.728854. eCollection 2021. PMID 34540697